CLINICAL TRIAL: NCT03220282
Title: Milk, Growth and Microbiota: A Randomized, Controlled Trial (RCT) of Donor Milk vs. Formula to Supplement Breastfeeding Late Preterm Newborns
Brief Title: The Milk, Growth and Microbiota Study
Acronym: MGM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling due to COVID-related restrictions.
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-21587
Record Dates: First submitted 2017-07-07; First posted 2017-07-18 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Preterm Infant; Growth Delay; Microbial Colonization; Breastfeeding; Breast Milk Substitute Intolerance
MeSH Terms: conditions — Premature Birth; Communicable Diseases; Breast Feeding | interventions — Food, Formulated

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 arms
Who Masked: Outcomes Assessor
Masking Description: Participant, PI, enrolling nurse and clinical care team will not be blinded as to treatment assignment. Outcomes will be assessed by blinded investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donor milk (Active Comparator): Pasteurized donor breast milk
  Interventions: Other: Donor milk
- Preterm infant formula (Placebo Comparator): Preterm formula determined by clinical practice
  Interventions: Other: Preterm infant formula

INTERVENTIONS:
Other: Donor milk — For late preterm newborns who are breastfeeding and whose mothers are not making enough breast milk yet to meet their nutritional needs, the study will compare the intervention of banked donor breast milk with the control of preterm infant formula.
  Other Names: Donor breast milk
  Arms: Donor milk
Other: Preterm infant formula — Preterm formula determined by clinical practice
  Other Names: Formula
  Arms: Preterm infant formula

SUMMARY:
Late preterm infants, who are born at 34, 35 or 36 weeks gestation, often have difficulty feeding, establishing growth, and fighting off infection. Breastfeeding provides improved nutrition to help fight infection, in part because breast milk encourages the growth of healthy bacteria (microbiota) in the infant's intestine. However, when mothers give birth preterm, their breasts are usually not quite ready to make milk; it can take several days to have enough breast milk to match a baby's nutritional needs. If there is not yet enough breast milk, formula is often used. However, formula can interfere with the growth of healthy intestinal bacteria. An alternate nutritional option is donor milk from a certified milk bank, which is available in all neonatal intensive care units (NICUs) in San Francisco. However, no scientific studies have yet studied donor milk for late preterm infants, so currently all San Francisco NICUs (as well as the large majority of NICUs nationwide) reserve donor milk for infants born at <34 weeks. This study's investigators therefore propose the "Milk, Growth and Microbiota (MGM) Study," a randomized controlled trial to compare banked donor milk to formula for breastfeeding late preterm infants born in San Francisco. Once enrolled in MGM, infants will be randomly assigned to receive either formula or banked donor milk if they need additional nutrition until their mothers are making enough milk. After enrolling the babies, investigators will weigh them daily to assess their growth. The investigators will also collect infant bowel movements at baseline, 1 week and 1 month to determine whether donor milk vs. formula impacts the type of bacteria in the baby's intestine. If the study's results show that donor milk optimizes growth while helping establish healthy bacteria in the baby's intestine, donor milk might be postnatal strategy to bolster neonatal nutrition for late preterm infants.

DETAILED DESCRIPTION:
In the U.S., 8% of all births occur between 34 0/7 and 36 6/7 weeks gestation and are regarded as late preterm birth. Compared to term newborns, late preterm newborns have a much higher risk of morbidity and mortality, in part because of difficulty establishing feeding and growth. Breastfeeding optimizes the nutrition of these infants by supporting growth and establishing a healthy intestinal microbiota. However, maternal breast milk production is often delayed after preterm birth, which can hamper optimal growth. When this occurs, clinicians may use formula to supplement breastfeeding. However, formula alters neonatal intestinal microbiota and can impede some of the benefits of a human milk diet. Donor milk from a certified milk bank could possibly be used instead of formula for supplementation prior to the onset of copious maternal milk production. However, the use of banked donor milk has never been studied in late preterm infants. The aim of this proposal is to report the effects of banked donor milk vs. formula on growth and on intestinal microbiota among late preterm, breastfeeding newborns who require additional nutrition before copious maternal milk is available. This study's investigators therefore propose a randomized, controlled trial enrolling late preterm newborns. Newborns will be randomly assigned either to breastfeed with additional formula feedings, or to breastfeed with additional donor milk feedings. The study's outcomes will be: (1) growth (rate of weight change), and (2) intestinal microbiota. If the study finds that temporary use of donor milk supports growth and maintains healthy intestinal microbiota until copious maternal milk becomes available, temporary use of donor milk might be a postnatal strategy to bolster neonatal nutrition and optimize nutritional support and growth for late preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Late preterm newborns >=34 weeks and <37 weeks gestation
* Breastfeeding
* Clinical team plans to start supplementation

Exclusion Criteria:

* Mothers are producing copious breast milk
* Birth weight <2100gm
* Any maternal or infant contraindication to breastfeeding

Ages: 1 Hour to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Weight change | Between enrollment and 24 hours after enrollment
  Grams

SECONDARY OUTCOMES:
Bifidobacteria | 1 week and 1 month after enrollment
  Abundance
Lactobacillus | 1 week and 1 month after enrollment
  Abundance
Clostridium | 1 week and 1 month after enrollment
  Abundance
Weight change | Between enrollment and 48 hours after enrollment
  Grams
Weight change | Between enrollment and 7 days of age
  Grams

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flaherman, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
The final data set will include information on infant weight and intestinal microbiota, as well as data on other clinical and demographic variables. Once the study has concluded and the data has been de-identified, the investigators will share the de-identified data with other users who agree to a data sharing plan that limits use of the data to research purposes only, excludes any use of the data to identify individual participants and destroys the data once the proposed research has been completed.